CLINICAL TRIAL: NCT04583644
Title: Pilot Trial of Fetoscopic Endoluminal Tracheal Occlusion (FETO) in Severe Left Congenital Diaphragmatic Hernia (CDH)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hanmin Lee (Other)
Responsible Party: Sponsor-Investigator, Hanmin Lee, Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-20723
Record Dates: First submitted 2018-06-12; First posted 2020-10-12 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Congenital Diaphragmatic Hernia
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Device - FETO (Experimental): Fetoscopic Endoluminal Tracheal Occlusion (FETO) surgery and removal of balloon using the BALT GOLDBAL2 balloon and BALTACCIBDPE100 catheter.
  Interventions: Device: Fetoscopic Endoluminal Tracheal Occlusion Surgery

INTERVENTIONS:
Device: Fetoscopic Endoluminal Tracheal Occlusion Surgery — Fetoscopic Endoluminal Tracheal Occlusion (FETO) surgery will be completed at 27 weeks 0 days - 29 weeks 6 days gestation.
  Fetoscopic removal of the balloon occlusion will be performed at 34 weeks 0 days to 34 weeks 6 days gestation.

SUMMARY:
Despite advances in prenatal diagnosis and postnatal therapies, including ECMO (Extracorporeal Membrane Oxygenation), inhaled nitric oxide therapy, and ventilator strategies that minimize ventilator-induced lung injury, morbidity and mortality rates for babies with severe CDH remain high. The rationale for fetal therapy in severe CDH is to promote adequate lung growth for neonatal survival. Prenatal tracheal occlusion obstructs the normal egress of lung fluid during pulmonary development leading to increased lung tissue stretch, increased cell proliferation, and accelerated lung growth. The investigator's goal with this pilot study is to study the feasibility of implementing Fetoscopic Endoluminal Tracheal Occlusion (FETO) therapy in the most severe group of fetuses with left CDH (LHR O/E < 25%).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age 18 years and older
* Singleton pregnancy
* Normal fetal karyotype with confirmation by culture results. Results by fluorescence in situ hybridization (FISH) will be acceptable if the patient is > 26 weeks
* Isolated Left CDH with liver up
* Gestation age at enrollment prior to 29 wks plus 6 days
* SEVERE pulmonary hypoplasia with US LHR O/E < 25% (measured at 180 to 295 weeks) at the time of surgery
* Gestational age at FETO procedure 27 weeks 0 days to 29 weeks 6 days as determined by clinical information (LMP) and evaluation of first ultrasound
* Family meets psychosocial criteria
* Pre-authorization from third-party payor for fetal intervention OR the ability to self-pay for study treatment. For all patients without insurance or the means to pay for the procedure, an attempt will be made to obtain Medicaid. Insurers that have denied payment have noted that this remains an experimental procedure. As this is a feasibility study and not being offered as either standard of care or as a prospective randomized control trial to determine efficacy, the investigators do not feel that there is a breach of ethical standards.
* Informed consent

Exclusion Criteria:

* Failure to meet all inclusion criteria
* Patient < 18 years of age
* Multi-fetal pregnancy
* Rubber latex allergy
* Preterm labor, cervix shortened (< 15 mm at enrollment or within 24 hours of FETO balloon insertion procedure) or uterine anomaly strongly predisposing to preterm labor, placenta previa
* Family does not meet psychosocial criteria. Reasons for exclusion include: insufficient social support, inability to understand requirements of the study, inability to reside in or near San Francisco.
* Right sided CDH or bilateral CDH, isolated left sided with LHR O/E < 25% (measured at 180 to 295 weeks) as determined by ultrasound
* Additional fetal anomaly by ultrasound, MRI, or echocardiogram at the fetal treatment center. Exclude chromosomal abnormalities, associated anomalies recognized to alter survival prognosis (ie. CDH and congenital heart disease) or presence of an underlying genetic syndrome (ie. Fryns). No cases will be removed post hoc if abnormalities are discovered in the course of post-operative monitoring
* Maternal contraindication to fetoscopic surgery or severe maternal medical condition in pregnancy
* History of incompetent cervix with or without cerclage
* Placental abnormalities (previa, abruption, accrete) known at time of enrollment
* Maternal-fetal Rh isoimmunization, Kell sensitization or neonatal alloimmune thrombocytopenia affecting the current pregnancy
* Maternal HIV, Hepatitis-B, Hepatitis-C status positive because of the increased risk of transmission to the fetus during maternal-fetal surgery. If the patient's HIV or Hepatitis status is unknown, the patient must be tested and found to have negative results before enrollment
* Uterine anomaly such as large or multiple fibroids or mullerian duct abnormality
* There is no safe or technically feasible fetoscopic approach to balloon placement
* Participation in another intervention study that influences maternal and fetal morbidity and mortality or participation in this trial in a previous pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-10-02 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Number of effective placements of balloon to occlude trachea via fetoscopy | Between 27 and 29 weeks gestation
  Number of effective placements of balloon to occlude trachea via fetoscopy by performing Fetoscopic Endoluminal Tracheal Occlusion (FETO) in fetuses with severe left congenital diaphragmatic hernia (CDH), as defined by lung to head ratio (LHR) Observed/Expected < 25%

SECONDARY OUTCOMES:
Rate of fetal lung growth after FETO as measured by lung volume. | Between 27 and 34 weeks gestation
  Fetal lung growth as measured by lung volume.
Rate of fetal lung growth after FETO as measured by Lung to head circumference ratio | Between 27 and 34 weeks gestation
  Fetal lung growth as measured by Lung to head circumference ratio (LHR) measurements.
Determine survival rate of FETO patients | 6 months after birth
  Survival at 6 months after birth.

CONTACTS AND LOCATIONS:
Overall Officials: Hanmin Lee, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco Fetal Treatment Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harrison MR, Adzick NS, Flake AW, Jennings RW, Estes JM, MacGillivray TE, Chueh JT, Goldberg JD, Filly RA, Goldstein RB, et al. Correction of congenital diaphragmatic hernia in utero: VI. Hard-earned lessons. J Pediatr Surg. 1993 Oct;28(10):1411-7; discussion 1417-8. doi: 10.1016/s0022-3468(05)80338-0. PMID 8263712
- [Background] Harrison MR, Keller RL, Hawgood SB, Kitterman JA, Sandberg PL, Farmer DL, Lee H, Filly RA, Farrell JA, Albanese CT. A randomized trial of fetal endoscopic tracheal occlusion for severe fetal congenital diaphragmatic hernia. N Engl J Med. 2003 Nov 13;349(20):1916-24. doi: 10.1056/NEJMoa035005. PMID 14614166
- [Background] Jani JC, Nicolaides KH, Gratacos E, Vandecruys H, Deprest JA; FETO Task Group. Fetal lung-to-head ratio in the prediction of survival in severe left-sided diaphragmatic hernia treated by fetal endoscopic tracheal occlusion (FETO). Am J Obstet Gynecol. 2006 Dec;195(6):1646-50. doi: 10.1016/j.ajog.2006.04.004. Epub 2006 Jun 12. PMID 16769018
- [Background] Adzick NS, Harrison MR, Glick PL, Villa RL, Finkbeiner W. Experimental pulmonary hypoplasia and oligohydramnios: relative contributions of lung fluid and fetal breathing movements. J Pediatr Surg. 1984 Dec;19(6):658-65. doi: 10.1016/s0022-3468(84)80349-8. PMID 6520670
- [Background] Bealer JF, Skarsgard ED, Hedrick MH, Meuli M, VanderWall KJ, Flake AW, Adzick NS, Harrison MR. The 'PLUG' odyssey: adventures in experimental fetal tracheal occlusion. J Pediatr Surg. 1995 Feb;30(2):361-4; discussion 364-5. doi: 10.1016/0022-3468(95)90590-1. PMID 7738765
- [Background] Jani JC, Nicolaides KH, Gratacos E, Valencia CM, Done E, Martinez JM, Gucciardo L, Cruz R, Deprest JA. Severe diaphragmatic hernia treated by fetal endoscopic tracheal occlusion. Ultrasound Obstet Gynecol. 2009 Sep;34(3):304-10. doi: 10.1002/uog.6450. PMID 19658113
- [Background] Deprest J, De Coppi P. Antenatal management of isolated congenital diaphragmatic hernia today and tomorrow: ongoing collaborative research and development. Journal of Pediatric Surgery Lecture. J Pediatr Surg. 2012 Feb;47(2):282-90. doi: 10.1016/j.jpedsurg.2011.11.020. PMID 22325377
- [Background] Harrison MR, Adzick NS, Flake AW, VanderWall KJ, Bealer JF, Howell LJ, Farrell JA, Filly RA, Rosen MA, Sola A, Goldberg JD. Correction of congenital diaphragmatic hernia in utero VIII: Response of the hypoplastic lung to tracheal occlusion. J Pediatr Surg. 1996 Oct;31(10):1339-48. doi: 10.1016/s0022-3468(96)90824-6. PMID 8906657
- See also: UCSF Fetal Treatment Center website — http://fetus.ucsf.edu/